High-Dose Dual Therapy vs Standard Triple Therapy for Treatment-Naïve H. Pylori: A Prospective Randomized Control Trial in a Diverse Urban New York City Population

PI: Ilan S Weisberg NCT05342532

Document Date: 1-2-2019



Icahn School of Medicine at Mount Sinai Mount Sinai Beth Israel Mount Sinai Brooklyn The Mount Sinai Hospital Mount Sinai Queens New York Eye and Ear Infirmary of Mount Sinai Mount Sinai St. Luke's Mount Sinai West Program for the Protection of Human Subjects Institutional Review Boards Mount Sinai Health System One Gustave L. Levy Place, Box 1081 New York, NY 10029-6574 T 212-824-8200 F 212-876-6789 irb@mssm.edu icahn.mssm.edu/pphs

## Initial Application IRB-19-01590 Ilan Weisberg

#### **Table of Contents**

| 1. Summary - Title | 1 |
|-------------------------------------|----|
| 2. Summary - Setup | 2 |
| 3. Summary - Background | 4 |
| 4. Research Personnel | 6 |
| 5. Sites | 7 |
| 6. Subjects - Enrollment | 8 |
| 7. Subjects - Setting and Resources | 9 |
| 8. Subjects - Populations | 10 |
| 9. Subjects - Participation | 11 |
| 10. Subjects - Risk and Benefits | 12 |
| 11. Procedures - Narrative | 13 |
| 12. Procedures - Genetic Testing | 14 |
| 13. Procedures - Details | 15 |
| 14. Procedures - Instruments | 16 |
| 15. Procedures - Compensation | 17 |
| 16. Consent - Obtaining Consent | 18 |
| 17. Consent - Documents | 19 |
| 18. Data - Collection | 20 |
| 19. Data - HIPAA | 21 |
| 20. Data - Storage | 22 |
| 21. Data - Safety Monitoring | 23 |
| 22. Financial Administration | 24 |
| 23. Attachments | 25 |

## 1. Summary - Title

#### **Protocol Title**

High Dose Dual Therapy vs. Clarithromycin Triple Therapy for Treatment Naive H. pylori Infection in an Urban Population: A Prospective, Randomized Clinical Trial

**Principal Investigator** 

Ilan Weisberg

When the application is complete, it will be sent to the PI for submission When the application is complete, it will be sent to the PI for submission

Primary Department Medicine - Gastroenterology

When the application is complete, it will be sent to the PI for submission

Application Initiated By Kelsey Collins

#### **Lay Summary**

H. pylori is the most prevalent chronic bacterial infection affecting humans in the world. H.pylori eradication rates using clarithromycin triple therapy are decreasing in the USA due to clarithromycin resistance. High dose dual therapy, consistent only of a proton pump inhibitor (PPI) and amoxicillin, is proving to be an effective alternative with higher eradication rates.

The purpose of our study is to determine if high dose dual therapy is as efficacious as the current standard treatment regimen of clarithromycin triple therapy for patients with Helicobacter pylori infection. The study will be a randomized, prospective clinical trial which will measure H. pylori eradication rates in patients with treatment naïve infection with either clarithromycin triple therapy or high dose dual therapy. This randomized clinical trial is relevant given the rising incidence of clarithromycin resistance that is seen in urban populations.

This is a phase 4 study looking at relative effectiveness of two regimens endorsed by the American College of Gastroenterology that use FDA-approved medications to treat H. pylori bacterial infection of the stomach. It will be a randomized study with subjects enrolled in one of the two treatment arms. There is no placebo group. The study aims to enroll a total of 166 subjects. Participating subjects will complete two weeks of therapy followed by a breath test to check for H. pylori eradication 4 weeks later, with a total participation time of 6 weeks. All tests and procedures are considered standard practice and there is no experimental intervention. The study is simply assessing the relative efficacy of two endorsed treatment regimens in our unique patient population.

IF Number IF2411170

## 2. Summary - Setup

Funding Has Been Requested /

Obtained

**Application Type** 

Request to Rely on Mount Sinai IRB

Research Involves Prospective Study ONLY

Consenting Participants Yes
Requesting Waiver or Alteration No

of Informed Consent for Any

**Procedures** 

Humanitarian Use Device (HUD)
Used Exclusively in the Course of

**Medical Practice** 

Use of an Investigational Device to NEvaluate Its Safety or Effectiveness

Banking Specimens for Future

Research

No

No

No

No

Cancer Related Research that Requires Approval from the Protocol Review and Monitoring

Committee (PRMC).

Is this Cancer Related Research? Cancer Related Research is defined as research that has cancer endpoints or has a cancer population as part of or all of its targeted population. This includes protocols studying patients with cancer or those at risk for cancer.

Clinical Trial Yes

\* A prospective biomedical or behavioral research study of human subjects that is designed to answer specific questions about biomedical or behavioral interventions (drugs, treatments, devices, or new ways of using known drugs, treatments, or devices).

\* Used to determine whether new biomedical or behavioral interventions are safe, efficacious, and effective.

Drugs / Biologics

No

- \* Drugs / Biologics That Are Not a Part of Standard Practice
- \* Controlled Substances
- \* Drugs / Biologics Supplied by the Research Sponsor or Purchased with Study Funds

Ionizing Radiation for imaging or therapy, including X-Ray, Fluoroscopy, CT, Nuclear Medicine, PET andor Radiation Therapy:

\* Purely for standard of care:

\* In frequency or intensity that exceeds what is necessary for

No No

No

standard of care:

Hazardous Materials

- \* Viral Vectors
- \* Plasmids
- \* Bacterial Artificial Chromosomes
- \* Toxic Chemicals, Potentially Toxic Medications, Carcinogens \* Autologous Cell Lines

Request Use of Clinical Research No Unit Resources

## 3. Summary - Background

#### **Objectives**

Is utilizing high dose dual therapy in treatment naïve adults diagnosed with H. pylori as effective as clarithromycin triple therapy in H. pylori eradication? Based on this information, should high dose dual therapy become a more widely utilized initial treatment regimen? We aim to determine if high dose dual therapy has comparable eradication rates for H. pylori infection when compared to clarithromycin triple therapy, specifically among our diverse New York City population. We will also assess the demographics among the population enrolled and being treated. We will then compare our data to that of recently published data describing the efficacy of high dose dual therapy as first line therapy in the management of H. pylori infection. Our main objective is to determine if using high dose dual therapy is non-inferior to standard triple therapy.

#### **Background**

Helicobacter pylori (HP) infection, the most prevalent chronic bacterial infection in the world, is the leading cause of peptic ulcer disease, chronic gastritis, gastric adenocarcinoma, and gastric mucosal associated lymphoid tissue (MALT) lymphoma. Its prevalence has been reported to be > 50% globally and roughly 35% within the United States. HP is also notably more prevalent amongst African American, Hispanic Americans, Asian Americans, and patients of low socioeconomic status. Per American College of Gastroenterology (ACG) guidelines, testing for HP should be done in patients with uninvestigated dyspepsia under the age of 60 without alarm features, patients with active PUD or history of PUD, patients on chronic treatment with NSAID's, and prior gastric malignancies. Although invasive testing using endoscopy with biopsy may be warranted in some patients, less invasive methods are available. Both the urea breath test (UBT) and the stool antigen assay are widely used, and both have sensitivities and specificities averaged at 95%.

Traditionally, HP infections have been empirically treated with standard triple therapy which includes a proton pump inhibitor (PPI), amoxicillin, and clarithromycin (metronidazole in those with penicillin allergy). Although initially found to be efficacious with an eradication rate of 77.5% in 2007, this number has been declining due to rising rates of antimicrobial resistance, particularly to clarithromycin. A recent retrospective study published in 2016 by Park, et al. evaluated clarithromycin resistance in the USA via DNA sequencing and found the resistance rate to be 32.3%. Current ACG guidelines advise to avoid clarithromycin triple therapy among populations where clarithromycin resistance rates exceed 15% and in patients with prior macrolide exposure.

High dose dual therapy (HDDT), a specific regimen of interest, has become an effective alternative to standard triple therapy, especially in areas with clarithromycin-resistance. This two-drug regimen, consistent of only a PPI and amoxicillin, is supported as an alternative regimen by the ACG and has limited data supporting its use as first line therapy. Its favorable qualities include a much lower bacterial resistance rate to amoxicillin, increased function of amoxicillin at an increased intragastric pH, less overall antibiotic exposure, and decreased propagation of clarithromycin resistance. Current data pertaining to its efficacy is limited to small population sizes and amongst specific populations in Asia and Europe. A recent study by Yang, et al. in 2015 evaluated the efficacy of HDDT vs. clarithromycin triple therapy in Taiwan, and found the eradication rate to be 95.3% vs. 80.7%, respectively.

We propose to conduct a prospective study aimed to determine if high dose dual therapy is as effective at HP eradication when compared to clarithromycin triple therapy amongst our diverse urban population in New York City.

#### **Primary and Secondary Study Endpoints**

Primary Endpoint: Eradication rate of HP infection treated with HDDT vs. clarithromycin triple therapy

Secondary Endpoints: Patient compliance with treatment regimen, patient satisfaction with treatment regimen, symptom control (assess improvement in epigastric pain, nausea, vomiting) adverse effects, age, sex, ethnicity, and country of origin

Protocol Was Already Approved
by the Icahn School of Medicine at
Mount Sinai (ISMMS) Institutional
Review Board (IRB) Under a
Different Principal Investigator

# 4. Research Personnel

| Name/Department | Role/Status | Contact | Access | Signature<br>Authority | Phone | Email |
|---|---|---|---|---|---|---|
| Ilan Weisberg /<br>Medicine -<br>Gastroenterology | PI/ | Yes | SIGNAUTH | | 212-844-1755 | |
| Kelsey Collins /<br>Medicine | Co-Investigator / | Yes | SIGNAUTH | | | |
| Daniel Pang / Office of Clinical Research | Study Coordinator /<br>Staff (non MD) | Yes | SIGNAUTH | | 212-420-4528 | |
| Ray Dong / Medicine - Gastroenterology | Co-Investigator / | Yes | SIGNAUTH | | | |

## 5. Sites

Site Name Mount Sinai Beth Israel

Other External Site Name

**Contact Details** 

Approved 1

**Approval Document** 

Funded By Mount Sinai

Reviewed By Mount Sinai IRB

Other IRB

IRB-19-01590 Initial Application Ilan Weisberg

# 6. Subjects - Enrollment

Site Name Mount Sinai Beth Israel

Subjects To Be Enrolled

Total Number of Subjects to be Enrolled Across All Listed Sites Above (Auto Populated) 0


## 7. Subjects - Setting and Resources

Setting of Human Research Faculty Practice Associates

**Total Number of Subjects Needed** 

166

**To Complete Study** 

**Feasibility of Meeting Recruitment Goals** 

We do not foresee any barriers to recruitment with a relatively high incidence of H. pylori seen in our large, ethnically diverse population.

**Facilities To Be Used for Conducting Research** 

Mount Sinai Downtown Union Square, 10 Union Square East, New York, NY 10003- Gastroenterology and Hepatology Clinic

**Multi-Center Study** 

Yes

Mount Sinai Principal Investigator is Responsible for All Centers

Yes

Management of Multi-Center Study

Co-Investigators are routinely present at the study site and are able to coordinate subject recruitment and screening for the study.

**Community-Based Participant** 

No

Research Study

## PI must attest to the following.

<sup>\*</sup> Process is adequately described to ensure that all persons assisting with the trial are adequately informed about the protocol, the investigational product(s), and their trial-related duties and functions.

## 8. Subjects - Populations

#### Inclusion Criteria

- 1. Male or female subject aged 18 years and older
- 2. Clinical diagnosis of H. pylori based on urea breath test
- 3. Treatment naïve adults
- 4. Subject willing to participate in the study and willing to give informed consent
- 5. Subject willing to take treatment regimen
- 6. Subject willing to return to clinic one month after finishing treatment to complete a survey and repeat urea breath testing

#### **Exclusion Criteria**

- 1. Previous H. pylori treatment failure
- 2. Antibiotic exposure within the past 4 weeks of H. pylori diagnosis
- 3. Documented or reported penicillin allergy
- 4. Pregnancy or breastfeeding
- 5. History of active gastric or non-gastric malignancy
- 6. Severe illness requiring hospitalization during treatment period
- 7. Starting additional antibiotic while on treatment

Enrollment Restrictions Based Yes

Upon Gender, Pregnancy, Childbearing Potential, or Race

Justify Restriction(s)

Amoxicillin is generally not recommended for pregnant women due to possible association with cleft lip and cleft palate.

Age Range(s) 18 to 64 Years, 65 Years and Over

Targeted Population(s) Adults - Patients

#### Other Aspects that Could Increase Subjects Vulnerability

There is a risk of loss of private health information, but there are procedures in place to minimize this risk.

#### Safeguards to protect Subjects rights and welfare

Data will be stored in REDCap, a web application for building and managing online surveys and databases. Institutional safeguards (such as disclosure of financial interests, HIPAA/ GCP training) are in place to guarantee protection of subjects' rights and welfare.

## 9. Subjects - Participation

#### **Duration of an Individual Subjects Participation in the Study**

Participation in this research study is expected to last up to 6 weeks for completion of both 2 week treatment and eradication testing 4 weeks later.

#### **Duration Anticipated to Enroll All Study Subjects**

1 year

Estimated Date for the Investigators Within two years to Complete This Study

#### **Procedures for Subjects to Request Withdrawal**

Subjects may withdraw by contacting the PI or research staff. Subjects may withdraw permission for the use and disclosure of any of the subject's protected information for research, but must do so in writing to the Principal Investigator at the address on the first page. Even if subject withdraws permission, the Principal Investigator for the research study may still use the information that was already collected if that information is necessary to complete the research study.

#### Procedures for Investigator to Withdraw Subjects

The study doctor or the institution may stop subject's involvement in this research study at any time without their consent. This may be because the research study is being stopped, the instructions of the study team have not been followed, the investigator believes it is in the subject's best interest, or for any other reason. If data have been stored as part of the research study, they too can be destroyed without your consent.

Participants Will Be Recruited Yes

**Recruitment Method(s)**Clinical Practice, Records (e.g. Medical, Employment, School), Physician Referral

#### **How Participants Will Be Identified**

Researchers will identify patients with treatment-naïve H. pylori with use of the urea breath test, which is routinely offered at the clinic. Potential subjects will be consented on the day of testing. If the test is positive, the laboratory will notify the physician and then randomization for treatment will occur, with subjects randomized to receive either clarithromycin triple therapy or high dose dual therapy. In addition, the study officials may look at the subject's clinic record to confirm the test results.

Who Will Initially Approach Member of Primary Care Team, Treating

Potential Participants Physician
How Research Will Be Introduced to Participants

## All patients with suspected H. pylori will be introduced to this study by their clinician, and if agreeable, they will be

consented for the study prior to urea breath testing. Potential subjects will consist of those on the research teams' clinic panel. Only if the urea breath test is positive, and the patient is consented, will the subject be randomized to receive treatment according to this study.

#### **How Participants Will Be Screened**

Participants will be screened based on the inclusion and exclusion criteria. Medical records will be viewed by the study personnel.

## 10. Subjects - Risk and Benefits

#### **Risks to Subjects**

The risk of loss of private information. Physical risks including medication side effects including headaches, GI upset, vulvovaginal infection, all of which are temporary and can be reversed. There is risk for a false negative result during urea breath testing, especially if the participant is taking a proton-pump inhibitor, bismuth, or antibiotics. This risk is also increased if the subject has an active peptic ulcer bleed.

#### Description of Procedures Taken to Lessen the Probability or Magnitude of Risks

Data will be stored in REDCap, a mature, secure web application for building and managing online surveys and databases. Study staff are also trained to use their utmost discretion when handling subject's protected health information.

#### Provisions for Research Related Harm / Injury

If the subject believes that they have suffered an injury related to this research as a participant in this study, they will contact the Principal Investigator for medical treatment.

#### **Expected Direct Benefit to Subjects**

There is no direct benefit to subjectss participating in the study.

#### **Benefit to Society**

Information from this study may benefit other people diagnosed with treatment naïve H. pylori in this urban population in the future.

#### **Provisions to Protect the Privacy Interests of Subjects**

Consent will be obtained in the Pl's/ Co-l's offices at the time of the subject's visit prior to any study assessments/ procedures. The investigator will approach eligible potential subjects and explain the study in a private room, including the reasons why subjects are eligible, risks and benefits and the regimens to be evaluated. Subjects privacy interests are always considered from the time subjects are identified for recruitment until they have completed the study. Only research personnel involved in the conduct of this research will have access to identifiable information and will be communicating with subjects throughout the trial. When trying to get in contact with subjects through mail or telephone messages etc., the utmost discretion will be utilized.

#### **Economic Impact on Subjects**

We do not foresee any additional expenses that the subject might incur from participation in this study. They will be billed according to their insurance plans. The subjects' clinical care will remain the same, with all subjects receiving 1 of 2 established antibiotic regimens for treatment therapy.

### 11. Procedures - Narrative

#### **Description of the Study Design**

Subjects with a diagnosis of treatment naïve H. pylori (B96.81) will be randomized to receive either high dose dual therapy (HDDT) or clarithromycin triple therapy.

Subjects will then receive an electronic prescription for their respective assigned regimen along with a medication log to self-report drug compliance.

After completing their assigned regimen, subjects will be scheduled for a post-treatment visit after 4 weeks. At this visit, subjects will undergo repeat urea breath testing. They will also bring in their medication log, pill bottles so that compliance can be recorded by research staff, and also complete a patient satisfaction survey.

#### **Description of Procedures Being Performed**

Patient survey- post treatment survey to determine patient satisfaction and patient compliance.

#### Description of the Source Records that Will Be Used to Collect Data About Subjects

Data collected will be entered into the REDCap database.

#### Description of Data that Will Be Collected Including Long-Term Follow-Up

Demographic data such as age, gender, and ethnicity. Subject health information such as presence or absence of concomitant medications, method of initial H. pylori diagnosis, and results from the eradication testing after treatment. Will also obtain patient satisfaction survey and patient compliance survey.

Research Requires HIV Testing No

# 12. Procedures - Genetic Testing

Genetic Testing Will Be Performed No Guidance and Policies > Future Use Data Sharing and Genetic Research


## 13. Procedures - Details

Surveys or Interviews Yes

Type of Instruments Being Used Created By Research Team

#### **Description of Instruments Created By Research Team**

A survey will be conducted for each subject at the end of their respective treatment regimen to assess patient satisfaction, patient compliance, and any adverse effects. In addition, subjects will be given a medication log to fill out after each dose of medication is taken. The subject will be instructed to return the log to clinic on their follow-up visit 4 weeks after completing treatment.

Audio / Photo / Video Recording No

**Deception** No

Results of the Study Will Be Shared Yes with Subjects or Others

How the Results Will Be Shared

Results of the eradication testing will be shared with the subject and explained by a qualified clinician.

When the Results Will Be Shared

Results will be shared in person or via telephone encounter once results are available from the lab.

## 14. Procedures - Instruments

### **Instruments Created By Research Team**

Type Medication Log

Name HDDT Medication Log

**Upload** Patient Medication Log-Dual Therapy.docx

Type Medication Log

Name Triple Therapy Medication Log

**Upload** Patient Medication Log- triple therapy.docx

Type Patient Survey
Name Patient Survey

Upload Day14\_Patient Survey.pdf


# 15. Procedures - Compensation

Compensation for Participation No


## 16. Consent - Obtaining Consent

Consent Process Adult Consent

#### Where and When Consent Will Be Obtained

Consent will be obtained during the operating hours of the Gastroenterology and Hepatology Clinic at Mount Sinai Downtown Union Square.

#### **Waiting Period for Obtaining Consent**

No waiting period is required for this study as both medications are approved for use by ACG for H. pylori. All patients with newly diagnosed, treatment naïve H. pylori and who meet the inclusion and exclusion criteria are being approached to participate in this study. Subjects will be given as much time as they need to consider if they want to participate in the study.

SOP HRP-090 Informed Consent Yes
Process for Research Is Being
Used

PPHS Worksheets, Checklists and SOPs

Process to Document Consent in Will Use Standard Template

Writing

Non-English Speaking Participants Yes

Will Be Enrolled

What Languages Other Than English Will Be Used

Spanish, Simplified Chinese

What Process Will Be Used Long Form

The consent document must be translated into the language of the potential subject, and approved by the IRB, before you can go through the consent process with the non-English speaking person. If, after the project is approved, a short form consent process is needed, please see the PPHS policy and submit a modification.

## 17. Consent - Documents

#### **Consent Documents**

Type Informed Consent

Name H. pylori Informed Consent

Upload HP\_Informed

Consent\_20190530\_v1.0\_clean.updated.docx

**Type** Research Study Figure

Name Figure of H. pylori Research Study
Upload Figure of H. pylori Research Study.docx

**Consent Templates** 

#### 18. Data - Collection

Health Related Information Will Be Yes Viewed, Recorded, or Generated

#### Description of Health Information That Will Be Viewed, Recorded, or Generated

Under the HIPAA waiver, medical records will be reviewed to ensure the date of initial positive urea breath test, list of current medications, any history of allergies, history of recent antibiotic use within 4 weeks, history of H. pylori infection, pregnancy status, and known comorbidities. In addition, the medical record will be reviewed to evaluate repeat urea breath testing after treatment is completed.

Non-Health Related Information Will Yes Be Viewed or Recorded

#### Description of Non-Health Information That Will Be Viewed or Recorded

Name, MRN, ethnic background, address, phone number, email address, and dates directly related to individuals

HIV / AIDS Related Information Will No

Be Viewed or Recorded

Data That Will Be Viewed, Yes

Recorded, or Generated Contains ANY of the Following Directly Identifiable Information

Will Be Viewed Name, Medical Record Number, Address

by street location, Telephone number, All Elements of Dates for Dates Directly Related to an Individual (i.e., Birth Date, Admission Date, Discharge Date), Email

Address

Will Be Recorded Name, Medical Record Number, Address

by street location, Telephone number, All Elements of Dates for Dates Directly Related to an Individual (i.e., Birth Date, Admission Date, Discharge Date), Email

Address

**Data Collection Sheet** 

A Data Collection Sheet is required if you are either performing a retrospective review, or your study meets the category of exempt 4 research, or your study meets the category of expedited 5 research. Please upload it here.

**Data Collection Source(s)** Participant, Medical Chart (Paper or

Electronic)

#### 19. Data - HIPAA

Obtaining HIPAA Authorization No
Requesting Waiver or Alteration Waiver
Research Could Be Practicably No
Conducted Without Access to
and Use of Protected Health
Information (PHI)

#### Explanation Why Research Could Not Be Practicably Conducted Without Access to and Use of PHI

Each patient's PHI must be accessed in order to review each patient's medical history in a retrospective manner, prior to inclusion in the study. Information including urea breath test results, history of H. pylori infection, recent antibiotic usage, allergies to medications, pregnancy status, and current medication regimen must be confirmed via PHI. In addition, by participating in the study, there will be new health information that must be added to the patient's PHI.

# Explanation Why Research Could Not Be Practicably Conducted Without a Waiver or Alteration of Authorization

Data must be collected from medical charts and the shared electronic medical database at the clinic contains information to help identify potential candidates for the study,

#### How PHI Will Be Protected from Improper Use or Disclosure

PHI will be stored according to the guidelines set by the PPHS data security standards. No patient identifiers will be used.

PHI Will Be Destroyed at the Yes Earliest Opportunity Consistent with the Research

#### When and How PHI Will Be Destroyed

PHI will be archived in REDCap after data analysis has been completed.

PHI Will Be Shared No

## PI must attest to the following.

\* I assure that the protected health information (PHI) will not be disclosed to any other person or entity not listed on this form except where required by law or for the authorized oversight of this research project. If at any time I want to reuse this PHI for other purposes or disclose it to other individuals or entities I will seek approval from the IRB.

## 20. Data - Storage

#### Location Where Data Will Be Stored

Data will be entered into a REDCap database. How will the data be stored? Other

#### Specify How Data Will Be Stored

Data will be entered into a REDCap database by authorized research staff that are listed in the research personnel

**Research Personnel Responsible** 

Ilan Weisberg

**Accessing Data** Yes **Receipt or Transmission of Data** Yes Holding Code That Can Be Linked No

to Identity of Participants

Research Personnel Responsible for:

Kelsey Collins

Yes **Accessing Data Receipt or Transmission of Data** Yes **Holding Code That Can Be Linked** No

to Identity of Participants

Research Personnel Responsible for:

**Daniel Pang** 

**Accessing Data** Yes **Receipt or Transmission of Data** Yes No

Holding Code That Can Be Linked to Identity of Participants

Ray Dong

Research Personnel Responsible

for:

**Accessing Data** Yes Receipt or Transmission of Data Yes **Holding Code That Can Be Linked** No

to Identity of Participants

**Duration Data Will Be Stored** 

Data will be stored for 7 years after the completion of this study.

#### Steps That Will Be Taken to Secure the Data During Storage, Use, and Transmission

Data will only be stored on the REDCap database and can only be accessed by research staff that can access the Mount Sinai network. On top of that, research staff will have to be given permission by database administrator to gain access to this database.

#### Power Analysis/Data Analysis Plan (Including Any Statistical Procedures)

Data will be analyzed without any identifying information. We plan to utilize t-tests (for continuous, normally distributed variables), the non-parametric Mann-Whitney test (for non normally distributed variables) and the chisquare test (for categorical variables).

IRB-19-01590 Initial Application Ilan Weisberg

## 21. Data - Safety Monitoring

More Than the Minimum Data No Safety Monitoring Will Be Done

The following minimum requirements apply to all projects, including retrospective reviews of medical records, use of tissue samples, and many minimal risk studies, such as observational and survey research. Because these minimum requirements apply to all studies, a specific written DSMP will not usually be required for projects that do not pose greater than minimal risk to subjects. The MSSM PPHS may alter the required level of monitoring if appropriate.

For all projects, the principal investigator must have a plan to assure that data integrity will be maintained during its collection, storage and analysis. All research projects must adhere to MSSM recommendations on the storage of research data. Loss of data containing identifiable information is reportable to the IRB within 5 business days. Any problems concerning the consent process and any subject complaints should be monitored by the investigator. Reports of such problems must be made at least annually. The discretion of the protocol director will guide the need to report these problems immediately or more frequently.

The principal investigator is, typically, the monitoring entity for the minimum DSMP. When a principal investigator is not a faculty member, the supervising faculty member must be responsible for the data and safety monitoring aspect of the protocol.

Will the Research Include Data No Coordinating Center Activities?

#### 22. Financial Administration

This information will help the Financial Administration of Clinical Trials Services (FACTS) office determine whether a Medicare Coverage Analysis (MCA) is needed for the research study. If you have any questions while completing this form, please contact the FACTS office at (212) 731-7067 or FACTS@mssm.edu.

Clinical Research Study Category Investigator Initiated

#### Payment Options:

- \* Option 1: No protocol-required services will be billed to patients or third-party payers. Does Not Need MCA
- \* Option 2: Protocol-required services (i.e., routine care services) will be billed to patients or third-party payers. Must Have MCA
- \* Option 3: Study is initiated and federally funded by a Government Sponsored Cooperative Group who will only pay for services that are solely conducted for research purposes and other protocol-required services (i.e., routine care services) will be billed to patients or third-party payers. Billing Grid Only Required, NO MCA
- \* Option 4: Study involves only data collection and has no protocol-required clinical services. Does Not Need MCA
- \* Option 5: Study is not described in any of the above options. Please describe the study and specify whether External Sponsor (i.e., industry, government, or philanthropic source) and/or patient/third party payer will pay for protocol required services. MCA MAY Be Required

**Payment Option** 

Option 1

No MCA is needed per option selected above.

#### Payment Option 1:

- \* Option 1A: Department/collaborating departments will act as internal sponsor paying for all protocol-required services and no protocol-required services will be billed to patients or third party payers.
- \* Option 1B: Study involves protocol-required clinical services and an External Sponsor (i.e., industry, government, or philanthropic source) will pay for all protocol-required services.

**Payment Option 1** 

Option 1A

# 23. Attachments

| Туре | Name | Version | Status | Filename | Uploaded<br>Date | |
|---|---|---|---|---|---|---|
| Instruments | Patient Medication<br>Log-Dual<br>Therapy.docx | 1 | New | Patient Medication<br>Log-Dual<br>Therapy.docx | 01/25/2019 | |
| Instruments | Patient Medication<br>Log- triple<br>therapy.docx | 1 | New | Patient Medication<br>Log- triple<br>therapy.docx | 01/25/2019 | |
| Consent Documents | HP_Informed<br>Consent_20190121_v | 1<br>/1.0.docx | New | HP_Informed<br>Consent_20190530_ | 05/30/2019<br>v1.0_clean.uլ | odated.docx |
| Instruments | Patient Survey.pdf | 1 | New | Day14_Patient<br>Survey.pdf | 02/08/2019 | |